CLINICAL TRIAL: NCT05980104
Title: Virtual Single-Session "Empowered Relief" Class for Individuals with Marfan Syndrome and Related Conditions
Brief Title: Single-Session "Empowered Relief" Class for Marfan Syndrome and Related Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: The Marfan Foundation (Other)
Responsible Party: Principal Investigator, Beth Darnall, Director of Stanford Pain Relief Innovations Lab, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 68906
Record Dates: First submitted 2023-07-25; First posted 2023-08-07 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain; Marfan Syndrome; Vascular Ehlers-Danlos Syndrome; Loeys-Dietz Syndrome
MeSH Terms: conditions — Chronic Pain; Marfan Syndrome; Ehlers-Danlos Syndrome, Type IV; Loeys-Dietz Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 1-Session pain relief skills class (online Empowered Relief) (Experimental): Empowered Relief is a 2-hour one session pain relief skills intervention that is delivered to a group of patients by a certified instructor using a standardized treatment manual and electronic slide deck. Content includes completion of a pain survey, pain neuroscience education, information on pain and stress responses, experiential exercises, information on three core pain management skills, completion of a personalized plan for empowered relief, and receipt of a binaural app for daily use.
  Interventions: Behavioral: Empowered Relief

INTERVENTIONS:
Behavioral: Empowered Relief — The participants will attend an online pain relief skills intervention (Empowered Relief). The two-hour group session is delivered by a certified instructor and includes pain neuroscience education, 3 core pain management skills, experiential exercises, completion of a personalized plan for empowered relief. Participants download a binaural relaxation audio file for daily use.
  Other Names: 1-Session Pain Relief Skills Intervention

SUMMARY:
Empowered Relief (ER) is a 1-session pain relief skills intervention that is delivered in-person or online by certified clinicians to groups of patients with acute or chronic pain. Prior work in has shown ER efficacy for reducing chronic pain, pain-related distress, and other symptoms 6 months post-treatment. The purpose of this study is to conduct the first feasibility and early efficacy test of online ER (two hours total treatment time) delivered to individuals with Marfan syndrome, Vascular Ehlers-Danlos Syndrome, Loeys-Dietz Syndrome, and related conditions. Participants will be followed for 3 months via 5 follow-up surveys.

DETAILED DESCRIPTION:
The investigators will implement a single arm online feasibility and preliminary efficacy trial of a pain relief skills intervention "Empowered Relief" to reduce pain metrics for individuals with Marfan syndrome and related conditions. Completion of the brief post-treatment survey is a binary measure of treatment engagement; treatment feasibility and appraisal are assessed with three items (satisfaction, perceived utility, and likelihood to use skills learned). Electronic surveys will measure pain intensity and symptom status at: baseline, immediately post-treatment; at post-treatment week 2 and months 1, 2, and 3. The study primary endpoint is change in pain intensity or pain interference from baseline to 1 month follow-up (short-term efficacy).

Online delivery of evidence-based behavioral treatment for pain will greatly expand access to patients across the U.S. living with Marfan syndrome and related conditions and associated chronic pain. Results from this study will fill several critical gaps in evidence for pain care in this population. This study will provide a low-cost, low-risk, widely available and feasible protocol that may help address the needs of patients living with Marfan and related syndromes.

Aim 1: Test the feasibility of live, online group-based ER.

Hypothesis 1a: Outcome 1, participant ratings will be >80% for the 7-item treatment appraisal/satisfaction measure administered immediately after completion of ER.

Hypothesis 1b: Outcome 2, ER attendance will be >70%.

Aim 2 (preliminary efficacy): Reduce multi-primary outcomes (pain intensity or pain interference) and secondary outcomes at 3 month post-treatment.

Hypothesis 2a: Outcome 3, Improvement of pain intensity or pain interference from baseline to 3 month follow-up (multi-primary study endpoint).

Hypothesis 2b: Outcome 4, Improvement of 4 priority secondary outcomes (sleep disturbance, pain catastrophizing, pain bothersomeness, and anxiety) from baseline to 3 month follow-up.

Hypothesis 2c: Outcome 5, Improvement of other secondary outcomes (satisfaction with social roles and responsibilities, anger, fatigue, and depression) from baseline to 3 month follow-up. Patient outcomes will be longitudinally tracked after the intervention session for participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 18 years of age or older
* Marfan Syndrome, Vascular Ehlers-Danlos Syndrome, Loeys-Dietz Syndrome or related connective tissue disease and chronic pain
* English fluency
* Ability to adhere to and complete study protocols

Exclusion Criteria:

* Cognitive impairment, non-English speaking, or psychological factors that would preclude comprehension of material and/or full participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Number of participants registered for class | baseline
  Full registration for the online session (N=100)
Class Attendance | at treatment
  At least 70% attendance for the registered Empowered Relief online class
Treatment appraisal | immediately post-treatment
  7 items assess treatment appraisal/satisfaction using 7-point scales (0-6) where higher ratings represent greater appraisal/satisfaction with the treatment. The investigators hypothesize >=80% ratings for treatment appraisal/satisfaction rated immediately post-treatment.

SECONDARY OUTCOMES:
Pain Intensity | post-treatment month 3
  Group pre-post reductions at 3 months with the Patient Reported Outcomes Measurement Systems (PROMIS) Pain Intensity 1-item scale assessing average pain intensity for the past 7 days (0= "No pain" to 10= "Worst pain imaginable") where a higher score represents a greater degree of pain intensity.
Pain Catastrophizing | post-treatment month 3
  Group pre-post changes at 3 months with the Pain Catastrophizing 13-item scale quantifying an individual's pain experience (5 point scale where 0 = "Not at all" and 4 = "All the time"). Scores range from 0-52 with higher scores indicating higher levels of pain catastrophizing.

OTHER OUTCOMES:
Pain Intensity | post-treatment month 1
  Group pre-post reductions at 1 month with the Patient Reported Outcomes Measurement Outcomes System (PROMIS) Pain Intensity 1-item scale assessing average pain intensity for the past 7 days (0= "No pain" to 10= "Worst pain imaginable") where a higher score represents a greater degree of pain intensity.
Pain Catastrophizing | post-treatment month 1
  Group pre-post changes at 1 month with the Pain Catastrophizing 13-item scale quantifying an individual's pain experience. Reponses range from 0 = "Not at all" and 4 = "All the time". Scores range from 0-52 with higher scores indicating higher levels of pain catastrophizing.
Pain Interference | post-treatment month 3
  Group pre-post changes at 3 months with the Patient Reported Outcomes Measurement Outcomes System (PROMIS) Pain Interference 8-item scale assessing pain interference with life enjoyment, concentration, and daily activities over the past 7 days. Responses range from 1 = "Not at all" to 5 = "Very much" where higher scores represent a greater degree of pain interference.
Pain Interference | post-treatment month 1
  Group pre-post changes at 1 month with the Patient Reported Outcomes Measurement Outcomes System (PROMIS) Pain Interference 8-item scale assessing pain interference with life enjoyment, concentration, and daily activities over the past 7 days. Responses range from 1 = "Not at all" to 5 = "Very much" where higher scores represent a greater degree of pain interference.
Sleep Disturbance | post-treatment month 3
  Group pre-post changes at 3 months with the Patient Reported Outcomes Measurement Outcomes System (PROMIS) Sleep Disturbance 6-item scale assessing sleep quality over the past 7 days. Responses range from 1 to 5 where higher scores represent lower sleep quality.
Sleep Disturbance | post-treatment month 1
  Group pre-post changes at 1 month with the Patient Reported Outcomes Measurement Outcomes System (PROMIS) Sleep Disturbance 6-item scale assessing sleep quality over the past 7 days. Responses range from 1 to 5 where higher scores represent lower sleep quality.
Pain Bothersomeness | post-treatment month 3
  Group pre-post changes at 3 months with the Pain Bothersomeness 1-item scale assessing pain bothersomeness over the past 7 days. Responses range from 0 = "Not at all bothersome" to 10 = "Extremely bothersome" where higher scores represent a greater degree of pain bothersomeness.
Pain Bothersomeness | post-treatment month 1
  Group pre-post changes at 1 month with the Pain Bothersomeness 1-item scale assessing pain bothersomeness over the past 7 days. Responses range from 0 = "Not at all bothersome" to 10 = "Extremely bothersome" where higher scores represent a greater degree of pain bothersomeness.
Fatigue | post-treatment month 3
  Group pre-post changes at 3 months with the Patient Reported Outcomes Measurement Outcomes System (PROMIS) Fatigue 8-item scale assessing fatigue over the past 7 days. Responses range from 1 = "Not at all" and "Never" to 5 = "Very much" and "Always" where higher scores represent a greater degree of fatigue.
Fatigue | post-treatment month 1
  Group pre-post changes at 1 month with the Patient Reported Outcomes Measurement Outcomes System (PROMIS) Fatigue 8-item scale assessing fatigue over the past 7 days. Responses range from 1 = "Not at all" and "Never" to 5 = "Very much" and "Always" where higher scores represent a greater degree of fatigue.
Satisfaction with Participation in Social Roles | post-treatment month 3
  Group pre-post changes at 3 months with the Patient Reported Outcomes Measurement Outcomes System (PROMIS) Satisfaction with Participation in Social Roles 7-item scale assessing satisfaction with performing one's usual social roles and activities. Responses range from 1 = "Not at all" to 5 "Very much" where higher scores represent greater satisfaction.
Satisfaction with Participation in Social Roles | post-treatment month 1
  Group pre-post changes at 1 month with the Patient Reported Outcomes Measurement Outcomes System (PROMIS) Satisfaction with Participation in Social Roles 7-item scale assessing satisfaction with performing one's usual social roles and activities. Responses range from 1 = "Not at all" to 5 "Very much" where higher scores represent greater satisfaction.
Pain Self-Efficacy Questionnaire | post-treatment month 3
  Group pre-post changes at 3 months with the Pain Self-Efficacy Questionnaire 2-item scale assessing confidence in functioning in the presence of pain. Responses range from 0 = "Not at all confident" to 6 = "Completely confident" where higher scores represent greater confidence in functioning.
Pain Self-Efficacy Questionnaire | post-treatment month 1
  Group pre-post changes at 1 month with the Pain Self-Efficacy 2-item scale assessing confidence in functioning in the presence of pain. Responses range from 0 = "Not at all confident" to 6 = "Completely confident" where higher scores represent greater confidence in functioning.
Depression | post-treatment month 3
  Group pre-post changes at 3 month with the Patient Reported Outcomes Measurement Outcomes System (PROMIS) Depression 6-item scale assessing negative mood in the past 7 days. Responses range from 1 = "Never" to 5 = "Always" where higher scores represent greater degree of depression.
Depression | post-treatment month 1
  Group pre-post changes at 1 month with the Patient Reported Outcomes Measurement Outcomes System (PROMIS) Depression 6-item scale assessing negative mood in the past 7 days. Responses range from 1 = "Never" to 5 = "Always" where higher scores represent greater degree of depression.
Anxiety | post-treatment month 3
  Group pre-post changes at 3 months with the Patient Reported Outcomes Measurement Outcomes System (PROMIS) Anxiety 6-item scale assessing fearfulness, worry and nervousness in the past 7 days. Responses range from 1 = "Never" to 5 = "Always" where higher scores represent greater degree of anxiety.
Anxiety | post-treatment month 1
  Group pre-post changes at 1 month with the Patient Reported Outcomes Measurement Outcomes System (PROMIS) Anxiety 6-item scale assessing fearfulness, worry and nervousness in the past 7 days. Responses range from 1 = "Never" to 5 = "Always" where higher scores represent greater degree of anxiety.
Anger | post-treatment month 1
  Anger: Within-subject baseline to 1 month the Patient Reported Outcomes Measurement Information System (PROMIS) Anger 5-item scale assesses anger over the past 7 days. Responses range from 1 = "Never" to 5 = "Always" where higher scores represent a greater degree of anger.
Anger | post-treatment month 3
  Anger: Within-subject baseline to 1 month the Patient Reported Outcomes Measurement Information System (PROMIS) Anger 5-item scale assesses anger over the past 7 days. Responses range from 1 = "Never" to 5 = "Always" where higher scores represent a greater degree of anger.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Darnall, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No